CLINICAL TRIAL: NCT04677829
Title: Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple-ascending-dose Trial to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacokinetics of Intravenous PNT001 in Hospitalized Patients With Traumatic Brain Injury (TBI)
Brief Title: Safety and Tolerability of PNT001 in Patients With Acute Traumatic Brain Injury (TBI)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to administrative, non-safety related reasons.
Sponsor: Pinteon Therapeutics, Inc (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PNT001-002
Record Dates: First submitted 2020-12-06; First posted 2020-12-21 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Escalating dose level cohorts; each cohort with an active and a placebo arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug will be administered and assessed in double-blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PNT001 1000mg (Experimental): PNT001 diluted in 5% dextrose for infusion
  Interventions: Biological: PNT001
- PNT001 4000mg (Experimental): PNT001 diluted in 5% dextrose for infusion
  Interventions: Biological: %5 dextrose for infusion
- Placebo (Placebo Comparator): 5% dextrose for infusion
  Interventions: Biological: PNT001; Biological: %5 dextrose for infusion

INTERVENTIONS:
Biological: PNT001 — 30 minute infusion for PNT001 1000mg; 60 minute infusion for PNT001 4000mg
  Arms: PNT001 1000mg; Placebo
Biological: %5 dextrose for infusion — 30 min placebo infusion for 1000mg; 60 minute placebo infusion for 4000mg
  Arms: PNT001 4000mg; Placebo

SUMMARY:
This is a Phase 1, multi-center, randomized, double-blind, placebo-controlled, multiple-ascending- dose trial to evaluate the safety, tolerability, immunogenicity, and pharmacokinetics of intravenous PNT001 in hospitalized patients with traumatic brain injury.

DETAILED DESCRIPTION:
The Phase 1 study is a double-blind, multiple ascending dose trial evaluating a total of 64 patients across two dose cohort groups. Each cohort will include 32 patients (24 active; 8 placebo) who will be randomized to receive three doses of either PNT001 or placebo. Doses studied will be 1000mg and 4000mg.

Patients admitted to the trauma center who meet entrance criteria will receive their first dose of study drug within 24 hours of documented TBI. They will remain in the facility for at least 24 hours after initial dose. Baseline biomarker collection and cognitive assessments will be completed. Study medication will be administered as an IV infusion over 30 minutes (for 1000mg cohort) or 60 minutes (for 4000mg cohort) followed by collection of safety, tolerability, pharmacokinetic, biomarker, imaging, and cognitive data over 12 weeks. Subsequent dosing visits will be at Days 28 and 56. All visits after initial discharge will be on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization due to documented evidence of TBI with Glasgow Coma Scale (GCS) Score 9-12 or GCS score of 13-15 with radiographic evidence of trauma.
2. Duration from documented time of TBI event to time of start of initial dose of study drug will not exceed 24 hours.
3. Signed informed consent by patient, or where applicable, patient's legally authorized representative.
4. Male and females, 18- 65 years of age at time of screening (State's legal age of majority is minimum age if higher than 18).
5. Female patients must meet protocol defined criteria for 1) non-childbearing potential, 2) post menopausal or 3) must have a negative pregnancy test and agree to contraception as outlined in the protocol.
6. Male must agree to use acceptable contraception and refrain from sperm donation during the entire study and for 200 days after dosing has been completed.
7. Has not participated in a clinical drug trial within 3 months of study start.
8. Body Mass Index (BMI) of 18.5-35.0 kg/m2 and for the 4000mg dose group only, weight greater than or equal to 44.8 kg.
9. Vision, hearing, speech, motor function, and comprehension sufficient for compliance with all testing procedures and assessments.

Exclusion Criteria:

1. TBI that does not require hospitalization.
2. TBI outside 24-hour window.
3. GCS < 9 within 2 hours of dosing.
4. History of TBI in past 12 months that resulted in patient seeking medical attention.
5. Evidence of penetrating head trauma or depressed skull fracture.
6. Clinical or radiographic evidence of mass effect, midline shift, or intracranial hypertension, requiring craniotomy/craniectomy.
7. Evidence of symptomatic cervical, thoracic, lumbar spine injury e.g. paresis, radiculopathy, that can be localized to the injury.
8. Systemic traumatic injury that would preclude participation in study or is expected to result in long-term disability.
9. Any other acute or chronic medical illness that in the judgement of the study physician results in functional impairment or impairs neuropsychiatric function.
10. Any acute intoxication that in the judgement of the study physician results in significant functional impairment or impairs neuropsychiatric function.
11. Any history of cancer within 5 years of enrollment with the exception of resected skin basal cell carcinoma.
12. Any major surgery requiring general anesthesia within 4 weeks of study drug administration.
13. Donation of blood or serum ≥500 mL to a blood bank or in a clinical study (except screening visit) within 3 months of study drug administration.
14. Known recent (within 6 months of study drug administration) drug or alcohol abuse as defined in DSM V, Diagnostic Criteria for Drug and Alcohol Abuse.
15. Evidence of any clinically significant neurological or psychiatric disorder that could interfere with study assessments as determined by investigator and sponsor.
16. Patient has history or currently has schizophrenia, schizoaffective disorder or bipolar disorder, untreated major depression (DSM-V or ICD-10 criteria).
17. Significant illness within the prior 30 days.
18. Abnormalities in creatinine, hepatic transaminases, or QT that would preclude entry into the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | 84 day study duration
  assess adverse events
Incidence of Treatment Emergent Clinical Laboratory Test Abnormalities | 84 day study duration
  measure clinical laboratory values
Incidence of Treatment Emergent Abnormalities in Physical Examination Findings | 84 day study duration
  perform physical examination
Incidence of Treatment Emergent Abnormalities in Neurological Examination Findings | 84 day study duration
  perform neurological examination
Incidence of Treatment Emergent Abnormalities in Vital Signs | 84 day study duration
  assess blood pressure, pulse, temperature, respiratory rate
Incidence of Treatment Emergent Abnormalities in 12-lead Electrocardiogram Assessment | 84 day duration of study
  measure ECG parameters

SECONDARY OUTCOMES:
Pharmacokinetic Properties of PNT001 in Serum | 84 day duration of study
  measure concentration of PNT001 in serum

OTHER OUTCOMES:
Anti-Drug Antibodies (ADA) | 84 day duration of study
  number of participants with presence of anti-drug antibodies (ADA) in serum
Biomarker Measurements in Plasma | 84 day duration of study
  measure concentrations of total (mid-domain) tau, NfL, GFAP, UCH-L1, pT181 tau, pT231 tau total tau in plasma
Effects of PNT001 on imaging parameters | Day 3 through the remainder of the 84 day study
  measure diffusion tensor imaging parameters
Effects of PNT001 on cognitive measures | 84 day duration of study
  scores on the Trails A and B assessments
Effects of PNT001 on health related Quality of Life | 84 day duration of the study
  measure change in ratings across 8 categories on the NeuroQOL assessment
Effects of PNT001 on a Global Outcome Scale | 84 day duration of the study
  measure disability outcome based on ratings in 8 areas of the Global Outcome Scale Extended (GOSE)
hsCRP Measurement in Serum | 84 day duration of the study
  measure concentrations of hsCRP in serum

CONTACTS AND LOCATIONS:
Overall Officials: Larry Altstiel, MD, PhD, Study Director — Pinteon Therapeutics
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No